CLINICAL TRIAL: NCT01177033
Title: ABC-Trial - Angioplasty or Bypass Surgery in Intermittent Claudication:
Brief Title: Angioplasty or Bypass Surgery in Intermittent Claudication
Acronym: ABC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut für Klinisch-Kardiovaskuläre Forschung GmbH (Network)
Collaborators: Technical University of Munich (Other)
Responsible Party: Univ.-Prof. Dr. Hans-Henning Eckstein, Klinikum Rechts der Isar, Technische Universität München
Other Study IDs: ISRCTN 39997806; 2010-021374-10 (EudraCT Number)
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2010-05

CONDITIONS: Intermittent Claudication; Complex Lesions of the Superficial Femoral Artery
MeSH Terms: conditions — Intermittent Claudication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Best endovascular treatment: Intervention type I: Best endovascular treatment (stent-protected angioplasty). Intervention type II: Best surgical treatment (femoro-popliteal bypass above the knee with autologous vein (1° choice) or a prosthetic graft (if vein is not available).
  Interventions: Other: Best endovascular treatment or Best surgical treatment
- Best surgical treatment: Intervention type I: Best endovascular treatment (stent-protected angioplasty). Intervention type II: Best surgical treatment (femoro-popliteal bypass above the knee with autologous vein (1° choice) or a prosthetic graft (if vein is not available).
  Interventions: Other: Best endovascular treatment or Best surgical treatment

INTERVENTIONS:
Other: Best endovascular treatment or Best surgical treatment — Intervention type I: Best endovascular treatment (stent-protected angioplasty). Intervention type II: Best surgical treatment (femoro-popliteal bypass above the knee with autologous vein (1° choice) or a prosthetic graft (if vein is not available).

SUMMARY:
CLINICAL TRIAL PROTOCOL SUMMARY / SYNOPSIS

Phase: IV

TITLE OF STUDY

Angioplasty or Bypass Surgery in Intermittent Claudication (ABC-Trial): a randomised controlled trial for patients with complex lesions of the superficial femoral artery

CONDITION

Peripheral arterial occlusive disease (PAOD)

OBJECTIVE(S)

The objective of this study is to evaluate the safety and efficacy of two therapeutic strategies (operative versus endovascular) in the treatment of patients with complex atherosclerotic lesions of the superficial femoral artery.

INTERVENTIONS

Intervention type I: Best endovascular treatment (stent-protected angioplasty). Intervention type II: Best surgical treatment (femoro-popliteal bypass above the knee with autologous vein (1° choice) or a prosthetic graft (if vein is not available).

Duration of intervention per patient: Dependent on the method of treatment

Follow-up per patient: 24 months

OUTCOMES

Primary efficacy endpoint:

Two primary efficacy endpoints will be considered simultaneously in this trial:

(A) Event-free survival (time-to-event endpoint): Proportion (over the course of time) of surviving patients who show a continuing clinical improvement of >= 1 class (Rutherford classification) without the need for repeated target lesion revascularization (TLR).

(B) Proportion of surviving patients with clinical improvement of >= 1 class (Rutherford classification) at 24 months after primary intervention (regardless any performed re-intervention).

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to verbally acknowledge and understanding of the associated risks, benefits, and treatment alternatives to therapeutic options of this trial. The patients, by providing informed consent, agree to these risks and benefits as stated in the patient informed consent document.
* Patients who are mentally and linguistically able to understand the aim of the study and to show sufficient compliance in following the study protocol.
* Age ≥ 50 and ≤ 85 years old.
* Intermittent claudication (IC) class 2 or 3 (Rutherford) assessed by treadmill testing or 6-Minute Walk Test.
* Lasting >3 months.
* Failed conservative therapy and the patient's desire for further treatment.
* Atherosclerotic single or multiple stenoses (>50%) or an occlusion of the Superficial Femoral Artery (SFA) with a target lesion length of 10-20 cm without involvement of the common/deep femoral artery and/or the popliteal artery confirmed by duplex ultrasound and angiography.
* At least one patent tibioperoneal artery with no stenosis >50% in diameter. Technical and morphological accessibility for both catheter intervention and bypass surgery.
* Absence of other disease that would limit exercise (e.g. angina or chronic respiratory disease).

Exclusion Criteria:

* >50% stenosis or occlusion of the iliac, the common, the deep femoral or the popliteal artery.
* Surgical reconstruction or catheter intervention on the index leg within the last six months.
* Unsuitability of treadmill testing / Six-Minute Walk Test. Chronic limb ischemia (intermittent claudication class 2 to 6) on the contralateral leg.
* Known allergy to contrast agents containing iodine.
* Contraindication for antiplatelet agents or anticoagulants.
* Clinically manifested heart insufficiency (NYHA III, IV) and/or uncorrected hyperthyreosis.
* Serious general disease state with an estimated life expectancy < 2 years (ASA IV, V).
* Pregnancy

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Intermittent Claudication, due to complex lesions of the superficial femoral artery
Sampling Method: Probability Sample
Enrollment: 470 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-08 (Estimated); Study Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (25):
- Austria (2):
  - Medizinische Universität Innsbruck, Innsbruck
  - Wilhelminenhospital Wien, Vienna
- Germany (23):
  - Universitätsklinikum Aachen, Aachen
  - Klinikum Augsburg, Augsburg
  - Klinikum am Bruderwald, Bamberg
  - Bundeswehrkrankenhaus Berlin, Berlin
  - Uniklinik Bonn, Bonn
  - Klinikum und Fachbereich Medizin Johann Wolfgang Goethe Universität Frankfurt am Main, Frankfurt am Main
  - Universitätsherzzentrum / Klinik und Poliklinik für Gefäßmedizin, Hamburg
  - Klinikum Hanau, Hanau
  - Universitätsklinikum Heidelberg, Heidelberg
  - Klinikum Ingolstadt, Ingolstadt
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - Klinikum Ludwigsburg, Ludwigsburg
  - Klinikum der Johannes Gutenberg Unviersität Mainz, Mainz
  - Universitätsklinikum Mannheim, Mannheim
  - Evangelisches Krankenhaus Mühlheim, Mühlheim
  - Klinikum der Universität München, Chirurgische Klinik und Poliklinik Innenstadt, München
  - Klinikum Rechts der Isar, Technische Universität München, München
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Regensburg, Regensburg
  - Diakonissen-Stiftungs-Krankenhaus Speyer, Speyer
  - Katharinenhospital Stuttgart, Stuttgart
  - Universtitätsklinikum Ulm, Ulm
  - HSK Dr. Horst Schmidt Klinik, Wiesbaden